CLINICAL TRIAL: NCT06139874
Title: Promoting Emotional Development Among Young Children Facing Adversity: An Effectiveness Implementation Study in St. Louis Schools
Brief Title: Thrive Intervention in Schools
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Joan Luby, MD, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202306092
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Childhood Mental Disorder
Keywords: Preschool; Parent-Child Relationship; Emotion Development; Therapy; Prevention
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Nicotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- THRIVE Coached (Experimental): Thrive is a promising early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention. It will be delivered by school social workers/counselors. Following training in THRIVE, school therapists in this condition will receive ongoing weekly group supervision over the life of the study.
  Interventions: Behavioral: THRIVE
- THRIVE Low Coached (Experimental): Thrive is a promising early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention. It will be delivered by school social workers/counselors. Following training in THRIVE, school therapists in this condition will receive weekly group supervision only during thier first THRIVE case.
  Interventions: Behavioral: THRIVE
- Parenting Wisely (Active Comparator): Online asynchronous parenting training that parents will complete independently.
  Interventions: Behavioral: Parenting Wisely

INTERVENTIONS:
Behavioral: THRIVE — Early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention.
  Arms: THRIVE Coached; THRIVE Low Coached
Behavioral: Parenting Wisely — Online asynchronous parenting program.
  Arms: Parenting Wisely

SUMMARY:
This study is designed to test the effectiveness and implementation of an early intervention therapy for children and their primary caregivers by using existing school counselors across several school districts.

The intervention is a 6-8 week caregiver-child intervention (THRIVE) which will be conducted via video conference in the family's home (i.e., zoom), or within the school setting (or a combination of those 2 modalities depending upon feasibility for the family). THRIVE will be compared to an asynchronous on-line parenting education program, Parenting Wisely (PW). This online parenting course will be accessed at www.parentingwisely.com.

Existing school counselors will be trained in the delivery of THRIVE to 3-7 year old children (in preschool, kindergarten and first grade) and their primary caregivers. In addition to testing the effectiveness of THRIVE compared to PW, we will also compare two implementation strategies: THRIVE-Coached and THRIVE-Low Coached (LC). We will assess ongoing coaching of THRIVE trainees to increase therapist efficacy and adherence to the intervention (THRIVE-Coached). This will be compared to implementation of THRIVE with low supports (e.g. weekly supervision) provided only for the first case following the initial training (THRIVE-LC].

Compared to those randomized to PW, we expect children who receive THRIVE will have significantly better behavioral and socio-emotional outcomes. Caregivers who receive THRIVE will experience less parenting stress and depression, more optimism and will show more nurturing, emotional tolerance, and supportive caregiving.

Therapists in the THRIVE-Coached condition will deliver the intervention with higher achieved outcomes and find the intervention to be more acceptable than therapists in the THRIVE-LC condition. Therapists in the THRIVE-Coached condition will be more likely to plan to sustain the intervention following the completion of the study than those in the THRIVE-LC condition. Parents and children receiving THRIVE from therapists in the THRIVE-Coached condition will have better socio-emotional outcomes than those in the THRIVE-LC and PW conditions.

ELIGIBILITY:
Inclusion Criteria:

* Near the clinical threshold on the Teacher or Parent Report Form
* An active primary caregiver can be identified and is available to participate in the intervention (mother, father, grandparent or any adult in this role)

Exclusion Criteria:

* Autism
* Major neurological disorder
* Participating in active weekly individual or family therapy

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 405 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2028-11-10 (Estimated); Study Completion 2028-11-10 (Estimated)

PRIMARY OUTCOMES:
Child Behavior Checklist | T1 (baseline), T2 (halfway through intervention), T3 (completion of intervention) and T4 (12 weeks post intervention)
  Measure of child psychopathology/impairment (emotional and behavioral functioning). Raw scores are converted into T-scores. The T-scores range from 50 to 100, with higher scores indicating more problematic behaviors. T-scores above 65 indicate psychiatric symptoms.

SECONDARY OUTCOMES:
The Emotion Regulation Checklist | T1 (baseline), T3 (completion of intervention)
  Measure of children's self-regulation that targets affective lability, intensity, valence, and flexibility. The total scores range from 24 to 96, with higher scores indicating better emotion regulation.
Coping with Children's Negative Emotions Scale | T1 (baseline), T2 (halfway through intervention), T3 (completion of intervention)
  Measure of parental coping styles in response to children's negative emotions. It consists of six subscales: Distress Reactions, Punitive Reactions, Expressive Encouragement, Emotion-Focused Reactions, Problem-Focused Reactions, and Minimization Reactions. The scores of each subscale range from 12 to 84, with higher scores indicating a greater likelihood of the parent engaging the type of response measured by that subscale.
Parenting Stress Index | T1 (baseline), T3 (completion of intervention)
  Measure of potential dysfunctional parent-child relationships and severity of parenting stress. Higher scores indicate higher levels of stress.
Parent-Child Observed Interaction Coding | T1 (baseline), T3 (completion of intervention)
  Objective ratings of the parent-child relationship functioning, parent emotion learning and child emotional competence.

OTHER OUTCOMES:
Beck Depression Inventory-II | T1 (baseline), T3 (completion of intervention)
  Measure of parental depression. The total scores range from 0 to 63, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Luby, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Early Emotional Development Program, St Louis, Missouri, United States

REFERENCES:
- See also: Early Emotional Development Program Website — http://eedp.wustl.edu/